CLINICAL TRIAL: NCT04336579
Title: Diaphragmatic Breathing Exercises As An Analgesia Adjunct in Total Knee Arthroplasty Patients in the Perioperative Period
Brief Title: Diaphragmatic Breathing Exercises in Total Knee Arthroplasty Patients
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Linda Rever, Clinical Associate Professor of Anesthesiology, University of Southern California
Other Study IDs: HS-19-00223
Record Dates: First submitted 2019-12-19; First posted 2020-04-07 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Anesthesia and Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Retrospective review of patients (participants) with standard analgesia post total knee arthroplasty
- Diaphragmatic Breathing: Intervention: Participants will perform diaphragmatic breathing exercises postoperatively as part of their multi-modal pain regimen.
  Interventions: Behavioral: Diaphragmatic Breathing

INTERVENTIONS:
Behavioral: Diaphragmatic Breathing — Simple diaphragmatic breathing exercise
  Groups: Diaphragmatic Breathing

SUMMARY:
Rationale: While total knee replacements (TKA) are one of the most commonly performed surgical procedures in the United States, this procedure can also be very painful. Postoperative mobilization and rehabilitation is vital to a patient's recovery, but inadequate pain control can impede patients' progress. Diaphragmatic breathing is an additional non-pharmacological and non-invasive tool with no adverse effects that could aid in recovery. This will serve as a pilot study for a possible larger controlled trials.

DETAILED DESCRIPTION:
Study population: Patients (participants) undergoing total knee arthroplasty at Keck USC Hospital at HC3

Study methodology: Patients (participants) will be taught with the aide of a handout and instructional videos preoperatively and in the recovery room on how to perform diaphragmatic breathing exercises for post-operative pain control. Patient (participant) pain levels will be assessed using the visual analog scale (VAS). The investigators will then be comparing VAS scores and daily opioid doses (morphine equivalents) between the study group and a control group. The control group will include prior patients (participants) over the past year who underwent TKA at Keck Hospital and also had pain scores and opioid usage measured, but did not receive the breathing treatment.

Study endpoints: Endpoints will include: pain levels via VAS scale, anxiety levels via VAS scale, and opioid usage (morphine equivalents).

ELIGIBILITY:
Inclusion Criteria:

* Patients (participants) undergoing total knee arthroplasty with a continuous peripheral nerve block catheter

Exclusion Criteria:

* Inability to perform or learn diaphragmatic breathing exercises or do not wish to participate in diaphragmatic breathing or study protocol
* Pregnant patients
* Patients without continuous peripheral nerve block catheter

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (participants) undergoing total knee arthroplasty with placement of continuous peripheral nerve block catheter between the ages of 50-90 years of age at the Keck Hospital of USC who want to participate and consent to participate in the study. The control group will be made up of patients( 50-90 years of age) who underwent total knee arthroplasty with placement of a continuous peripheral nerve block catheter over the year prior, without participation in breathing exercises, at the Keck Hospital of USC.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain Level | Prior to intervention
  Verbal Analog Pain Score - rate pain on 0-10 scale where 0=no pain, 10= worst possible pain
Opioid Usage (morphine equivalents) | Prior to intervention
  Opioid Usage for pain
Anxiety Level | Prior to intervention
  Verbal Analog Score -rate anxiety on 0-10 scale where 0= no anxiety, 10= worst possible anxiety
Pain Level | 15 minutes after intervention
  Verbal Analog Pain Score - rate pain on 0-10 scale where 0 =no pain, 10 = worst possible pain
Opioid Usage (morphine equivalents) | 15 minutes after intervention
  Opioid Usage for pain
Anxiety Level | 15 minutes after intervention
  Verbal Analog Score - rate anxiety on 0-10 scale where 0 =no anxiety, 10 = worst possible anxiety
Pain Level | 6 hours after intervention
  Verbal Analog Pain Score - rate pain on 0-10 scale where 0 =no pain, 10 = worst possible pain
Opioid Usage (morphine equivalents) | 6 hours after intervention
  Opioid Usage for pain
Anxiety Level | 6 hours after intervention
  Verbal Analog Score- rate anxiety on 0-10 scale where 0 =no anxiety, 10 = worst possible anxiety
Pain Level | 1 day after intervention
  Verbal Analog Pain Score - rate pain on 0-10 scale where 0 =no pain, 10 = worst possible pain
Opioid Usage (morphine equivalents) | 1 day after intervention
  Opioid Usage for pain
Anxiety Level | 1 day after intervention
  Verbal Analog Score - rate anxiety on 0-10 scale where 0 = no anxiety, 10 = worst possible pain

CONTACTS AND LOCATIONS:
Overall Officials: Linda J Rever, MD, Principal Investigator — University of Southern California
Locations (1):
- Keck Hospital of USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No